CLINICAL TRIAL: NCT02507622
Title: E-NOSE for Breath Gas Analysis Under Microgravity Conditions
Acronym: E-NOSE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 14-103
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Last update posted 2015-07-24 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gas concentration (Other): Gaz concentration of C02, CO and NH4, 3 exhaled in weightlessness and normal gravity.
  Interventions: Other: measurement of the concentration of C02, CO and NH4, 3 exhaled gas with E-Nose system; Other: Parabolic flight

INTERVENTIONS:
Other: measurement of the concentration of C02, CO and NH4, 3 exhaled gas with E-Nose system
Other: Parabolic flight

SUMMARY:
The main goal of the study is demonstrate that e-Nose system function is not altered in weightlessness and more specifically that gas concentration measurements are the same in weightlessness and normal gravity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (men or women)
* Aged from 20 to 65
* Affiliated to a French Social Security system or, for people living abroad, holding a European Health Insurance Card (EHIC)
* Who accepted to take part in the study
* Who has given their written stated consent
* Who has passed a medical examination similar to a standard aviation medical examination for private pilot aptitude (JAR FCL3 Class 2 medical examination). There will be no additional test performed for subject selection

Exclusion Criteria:

* Person who took part in a previous biomedical research protocol, of which exclusion period is not terminated
* Pregnant women

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2014-09; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
The judgment criteria are the concentration of C02, CO and NH4, 3 exhaled gas | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France